CLINICAL TRIAL: NCT05701007
Title: Real World Evidence Study on Metastatic Prostate Cancer Patient Characteristics, Treatment Patterns and Outcomes in the Pirkanmaa Hospital District in Finland
Brief Title: Real World Evidence Study on Metastatic Prostate Cancer in the Pirkanmaa Hospital District in Finland
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441057; PrCa-RWD (Other: Alias Study Number)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration Sensitive Prostate Cancer (mCSPC); Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: mCRPC; metastatic prostate cancer; registry study; RWE; real world evidence; Finland; Metastasis; Prostatic Neoplasms; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — abiraterone; enzalutamide; Docetaxel; apalutamide; cabazitaxel; Radium-223; Lutetium-177; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin; Leuprolide; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with metastatic castration sensitive prostate cancer (mCSPC)
  Interventions: Drug: degarelix; Drug: goserelin; Drug: leuprorelin; Drug: triptorelin
- Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
  Interventions: Drug: abiraterone; Drug: enzalutamide; Drug: docetaxel; Drug: apalutamide; Drug: cabazitaxel; Drug: Radium-223; Drug: Lutetium-177

INTERVENTIONS:
Drug: abiraterone — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: enzalutamide — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: docetaxel — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: apalutamide — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: cabazitaxel — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: Radium-223 — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: Lutetium-177 — mCRPC
  Groups: Patients diagnosed with metastatic castration resistant prostate cancer (mCRPC)
Drug: degarelix — mCSPC
  Groups: Patients diagnosed with metastatic castration sensitive prostate cancer (mCSPC)
Drug: goserelin — mCSPC
  Groups: Patients diagnosed with metastatic castration sensitive prostate cancer (mCSPC)
Drug: leuprorelin — mCSPC
  Groups: Patients diagnosed with metastatic castration sensitive prostate cancer (mCSPC)
Drug: triptorelin — mCSPC
  Groups: Patients diagnosed with metastatic castration sensitive prostate cancer (mCSPC)

SUMMARY:
Comprehensive understanding of the epidemiology and disease burden of metastatic prostate cancer patients in Finland is lacking. This study will address the following questions:

* What are the demographic and clinical characteristics of metastatic prostate cancer patients?
* How are metastatic prostate cancer patients currently treated and how effective are these treatments?
* How does the development of castration-resistance affect patient outcomes?
* What is the economic burden of metastatic prostate cancer?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer between 1/1/2007 - 12/31/2022
* Resident of Pirkanmaa at index date (diagnosis of mCSPC and/or mCRPC)
* Detection of metastatic prostate cancer

Exclusion Criteria:

* Prevalent mCSPC and mCRPC patients (mCSPC or mCRPC diagnosis date before 1/1/2014
* Patient has another cancer diagnosis or the patient has received chemotherapy other than docetaxel or cabazitaxel within 2 years of mPC diagnosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with cancer of the prostate.
Study Population: Adult patients with advanced/metastatic prostate cancer and medical records available in the Hospital District of Pirkanmaa, Finland registry
Sampling Method: Non-Probability Sample
Enrollment: 1083 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants aged >=18 years who were diagnosed with metastatic prostate cancer (mPC)- metastatic castration sensitive prostate cancer (mCSPC) and/or metastatic castration resistant prostate cancer (mCRPC) between 01-Jan-2014 and 31-Dec-2022 (approximately 9 years) were identified from Pirkanmaa Hospital District (PHD) data records and their data were included in this study.
Pre-assignment Details: Available data from eligible participants was evaluated in approximately 14 months (study start date: 13-Feb-2023 to study completion date:10-Apr-2024) of this retrospective, observational study as per its objectives.
Groups:
- Participants Diagnosed With mPC: Eligible participants with mPC and whose data were evaluated retrospectively.
Period: Overall Study
Arm/Group | Participants Diagnosed With mPC
Started | 1083
Participants Diagnosed With mCSPC | 795
Participants Diagnosed With mCRPC | 558
Completed | 1083
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants Diagnosed With mPC
Number analyzed (Participants) | 1083
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Participants were not exclusive in mCSPC and mCRPC cohorts.
  Years
    mCSPC: number analyzed (Participants) | 795
    mCSPC | 73.8 (9)
    mCRPC: number analyzed (Participants) | 558
    mCRPC | 75.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were not exclusive in mCSPC and mCRPC cohorts.
  Participants
    mCSPC: number analyzed (Participants) | 795
    mCSPC: Female | 0
    mCSPC: Male | 795
    mCRPC: number analyzed (Participants) | 558
    mCRPC: Female | 0
    mCRPC: Male | 558
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass. It is widely used as a general indicator of whether a participant has a healthy body weight for their height. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: 3 months before index date (closest value); retrospective available data evaluated in this study for approximately 14 months
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Analysis excluded participants with missing data.
Measure: Mean (Standard Deviation); unit: Kilogram per meter square
Groups:
- Participants Diagnosed With mCSPC: Eligible participants with mCSPC and whose data were evaluated retrospectively.
- Participants Diagnosed With mCRPC: Eligible participants with mCRPC and whose data were evaluated retrospectively.
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 228 | 149
Kilogram per meter square | 27.9 (12.4) | 27.1 (4.7)

2. Primary Outcome: Prostate-Specific Antigen (PSA)
Description: PSA is a protein produced by the prostate gland, and the PSA test measures its levels in the blood. It is primarily used to screen for prostate cancer and monitor participants after treatment. Elevated PSA levels may indicate prostate cancer or other prostate abnormalities. Common prostate abnormalities include benign prostatic hyperplasia, prostatitis, prostate cancer. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 487 | 514
Nanogram per milliliter | 199.7 (704.7) | 92 (396.4)

3. Primary Outcome: Alkaline Phosphatase (P-AFOS)
Description: Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 338 | 457
Units per liter | 214.1 (402.3) | 144 (221.8)

4. Primary Outcome: Length of Follow-up
Description: as for outcome 3
Time Frame: From index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Years | 1.8 (1.8) | 1.9 (1.6)

5. Primary Outcome: Number of Participants With de Novo Metastasis
Description: The new metastasis was defined based on the prostate cancer diagnosis dates within 2 months from the index date. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to metastatic castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered new CRPC).
Time Frame: Within 2 months from index date; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 444 | 240

6. Primary Outcome: Number of Participants Who Received Treatment for mCRPC and mCSPC
Description: Number of participants who received treatment for mCRPC and mCSPC were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: Post index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 668 | 536

7. Primary Outcome: Number of Participants Diagnosed With mCSPC Who Progressed to mCRPC
Description: Number of participants initially diagnosed With mCSPC who progressed into mCRPC were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Only reporting arm "Participants Diagnosed With mCSPC" is reported as this outcome measure was to be analyzed for participants who had mCSPC and they progressed to mCRPC.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC
Number analyzed (Participants) | 795
Participants | 270

8. Primary Outcome: Number of Participants With Orchiectomy
Description: Number of participants with orchiectomy done were reported in this outcome measure. Orchiectomy is a surgical procedure in which one or both testicles are removed. It is commonly performed to treat or prevent prostate cancer from spreading. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: Closest record any time from index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 10 | 9

9. Primary Outcome: Number of Participants Undergone Palliative Radiology
Description: Number of participants with palliative radiology done were reported in this outcome measure. This is a treatment designed to alleviate symptoms caused by advanced cancer, rather than cure the disease. It is commonly used to reduce tumor size or provide relief from pain, bleeding, or obstructions, ultimately enhancing the participant's quality of life. It is especially beneficial for participants with cancers that cannot be cured, offering relief from distressing symptoms such as tumor compression on organs or bones, as well as severe pain. Palliative radiology is analyzed based on procedure code (WF049). Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 222 | 187

10. Primary Outcome: Number of Participants With Symptomatic Skeletal-Related Event (SSRE)
Description: SSRE was defined as bone instability related to the treatment of advanced prostate cancer or due to the spread of prostate cancer to the bone (metastases). Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 44 | 43

11. Primary Outcome: Number of Participants With Osteoporosis
Description: Number of participants with osteoporosis were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 558 | 795
Participants | 9 | NA — According to the guidelines set by the Finnish Health and Social Data Permit Authority (Findata), results having less than 5 participants with events cannot be exported from Findata data servers due to participant privacy restrictions.

12. Primary Outcome: Number of Participants Who Were on Bone Medication
Description: Number of participants who were on bone medication (denosumab, zoledronic acid) were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 154 | 292

13. Primary Outcome: Number of Participants Who Were on Opioids
Description: Number of participants who were on opioids (morphine, oxycodone, fentanyl, methadone, hydromorphone) were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants | 310 | 332

14. Primary Outcome: Number of Participants Classified Per Charlson Comorbidity Index (CCI) Scores
Description: CCI score range was from 0 to 14, where 0= low comorbid condition and 14= high comorbid condition, higher scores indicated more comorbidity. CCI was reported based on comorbidities reported 5 years before the index (index date included). Participants with grade 4 or more than 4 were combined and presented to avoid risk of re-identification of participants. Only those categories are reported which had at least 1 participant data in any of the reporting group. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: Up to 5 years before the index date (index date included); retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants
  0 level | 548 | 329
  1 level | 147 | 142
  2 level | 61 | 52
  3 level | 25 | 25
  4+ level | 14 | 10

15. Primary Outcome: Number of Participants Classified Per Gleason Score
Description: Gleason score is used to grade tumors based upon its microscopic appearance. Gleason scores range from 1 (low-grade cancer) to 10 (high-grade cancer). Low grade prostate cancer grows more slowly than high-grade cancer and is less likely to spread (metastasize). Scores from 3-5 have been combined to avoid risk of re-identification of participants. Only those categories are reported which had at least 1 participant data in any of the reporting group. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: Closest record any time from index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx.9 years; retrospective available data evaluated in this study for approx.14 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Participants
  3-5 | 7 | 12
  6 | 46 | 31
  7 | 171 | 88
  8 | 100 | 71
  9 | 369 | 286
  10 | 48 | 40
  Missing | 54 | 30

16. Primary Outcome: Number of Participants Based on Tumor Node Metastasis (TNM) Classification: T
Description: T categories: T1, T2, T3, T4; In this, T describes the size of the tumor and any spread of cancer into nearby tissue. Numbers after the T (such as T1, T2, T3, and T4) describe tumor size and/or amount of spread into nearby structures. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC). Higher numbers indicate greater the tumor size.
Time Frame: Closest record during 3 months before or after the index date; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 178 | 70
Participants
  TNM (T): T1 | 13 | 0
  TNM (T): T1-T2 | 0 | 12
  TNM (T): T2 | 28 | 0
  TNM (T): T3 | 81 | 38
  TNM (T): T4 | 56 | 20

17. Primary Outcome: Number of Participants Based on Tumor Node Metastasis (TNM) Classification: N
Description: N categories: N0, N1, N2, NX. N describes spread of cancer to nearby lymph nodes. Numbers after the N (such as N0, N1, N2, NX) describe tumor size and/or amount of spread into nearby structures. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC). Higher numbers indicate greater the tumor size and spread into nearby lymph nodes.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 112 | 42
Participants
  TNM(N): N0 | 41 | 17
  TNM(N): N1 | 65 | 0
  TNM(N): N1-N2 | 0 | 25
  TNM(N): N2-N3 | 6 | 0

18. Primary Outcome: Number of Participants Based on Tumor Node Metastasis (TNM) Classification: M
Description: M categories: M0, M1. M describes metastasis (spread of cancer to other parts of the body). Numbers after the M (such as M0, M1) describe tumor size and/or amount of spread into nearby structures. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC). Higher numbers indicate greater the tumor size and spread into nearby body parts.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 163 | 65
Participants
  TNM(M): M0 | 50 | 29
  TNM(M): M1 | 113 | 36

19. Primary Outcome: Number of Participants Based on Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Description: ECOG PS is a scale to assess a participant's disease status. 0 = fully active, able to carry out all pre-disease performance without restriction; 1 = restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = ambulatory and capable of all self-care, unable to carry out any work activities. up and about > 50% of waking hours; 3 = capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = completely disabled, confined to bed or chair; 5 = dead. Only those categories are reported which had at least 1 participant data in any of the reporting group. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 469 | 303
Participants
  0 | 175 | 97
  1 | 181 | 112
  2 | 64 | 67
  3 | 38 | 0
  3-4 | 0 | 27
  4 | 11 | 0

20. Primary Outcome: Number of Participants According to Treatment Per Treatment Line for mPC: mCSPC Participants
Description: Number of participants according to treatment per treatment line (first, second, third and fourth line) for mPC for mCSPC participants were reported in this outcome measure. Palliative care was analyzed based on International Classification of Diseases- 10th revision (ICD-10) code Z51.5. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows. Only reporting arm "Participants Diagnosed With mCSPC" is reported as this outcome measure was planned to be analyzed for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC
Number analyzed (Participants) | 668
Participants
  First line: Palliative care | 60
  First line: Apalutamide | 8
  First line: Bicalutamide | 60
  First line: Degarelix | 244
  First line: Docetaxel | 39
  First line: Goserelin | 22
  First line: Leuprorelin | 175
  First line: Triptorelin | 31
  First line: Other | 5
  First Line: Unknown | 24
  Second line: Palliative care | 24
  Second line: Apalutamide | 21
  Second line: Bicalutamide | 42
  Second line: Degarelix | 21
  Second line: Docetaxel | 89
  Second line: Goserelin | 12
  Second line: Leuprorelin | 50
  Second line: Triptorelin | 18
  Second line: Other | 8
  Second Line: EOF | 140
  Second Line: Death | 98
  Second Line: Unknown | 145
  Third Line: Palliative care: number analyzed (Participants) | 285
  Third Line: Palliative care | 10
  Third Line: Apalutamide: number analyzed (Participants) | 285
  Third Line: Apalutamide | 7
  Third Line: Docetaxel: number analyzed (Participants) | 285
  Third Line: Docetaxel | 5
  Third Line: Leuprorelin: number analyzed (Participants) | 285
  Third Line: Leuprorelin | 17
  Third Line: Triptorelin: number analyzed (Participants) | 285
  Third Line: Triptorelin | 7
  Third Line: Other: number analyzed (Participants) | 285
  Third Line: Other | 12
  Third Line: EOF: number analyzed (Participants) | 285
  Third Line: EOF | 87
  Third Line: Death: number analyzed (Participants) | 285
  Third Line: Death | 36
  Third Line: Unknown: number analyzed (Participants) | 285
  Third Line: Unknown | 104
  Fourth Line: Palliative care/Unknown: number analyzed (Participants) | 58
  Fourth Line: Palliative care/Unknown | 21
  Fourth Line: EOF: number analyzed (Participants) | 58
  Fourth Line: EOF | 20
  Fourth Line: Death: number analyzed (Participants) | 58
  Fourth Line: Death | 11
  Fourth Line: Other: number analyzed (Participants) | 58
  Fourth Line: Other | 6

21. Primary Outcome: Number of Participants According to Treatment Per Treatment Line for mPC: mCRPC Participants
Description: Number of participants according to treatment per treatment line (first, second, third and, fourth, and fifth line) for mPC for mCRPC participants were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 6
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows. Only reporting arm "Participants Diagnosed With mCRPC" is reported as this outcome measure was planned to be analyzed for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 536
Participants
  First line: Palliative care | 23
  First line: Abiraterone | 77
  First line: Apalutamide | 5
  First line: Bicalutamide | 59
  First line: Degarelix | 23
  First line: Docetaxel | 55
  First line: Enzalutamide | 190
  First line: Flutamide | 10
  First line: Goserelin | 16
  First Line: Leuprorelin | 42
  First Line: Radium-223 | 11
  First Line: Other | 25
  Second line: Palliative care | 73
  Second line: Abiraterone | 65
  Second line: Bicalutamide | 22
  Second line: Cabazitaxel | 18
  Second line: Docetaxel | 37
  Second line: Enzalutamide | 90
  Second line: Flutamide | 15
  Second line: Radium-223 | 7
  Second line: Other | 10
  Second Line: EOF | 123
  Second Line: Death | 76
  Third Line: Palliative care: number analyzed (Participants) | 337
  Third Line: Palliative care | 59
  Third Line: Abiraterone: number analyzed (Participants) | 337
  Third Line: Abiraterone | 32
  Third Line: Bicalutamide: number analyzed (Participants) | 337
  Third Line: Bicalutamide | 5
  Third Line: Cabazitaxel: number analyzed (Participants) | 337
  Third Line: Cabazitaxel | 23
  Third Line: Docetaxel: number analyzed (Participants) | 337
  Third Line: Docetaxel | 16
  Third Line: Enzalutamide: number analyzed (Participants) | 337
  Third Line: Enzalutamide | 35
  Third Line: Radium-223: number analyzed (Participants) | 337
  Third Line: Radium-223 | 9
  Third Line: Other: number analyzed (Participants) | 337
  Third Line: Other | 5
  Third LIne: EOF: number analyzed (Participants) | 337
  Third LIne: EOF | 56
  Third Line: Death: number analyzed (Participants) | 337
  Third Line: Death | 97
  Fourth Line: Palliative care: number analyzed (Participants) | 184
  Fourth Line: Palliative care | 44
  Fourth Line: Abiraterone: number analyzed (Participants) | 184
  Fourth Line: Abiraterone | 13
  Fourth Line: Cabazitaxel: number analyzed (Participants) | 184
  Fourth Line: Cabazitaxel | 16
  Fourth Line: Docetaxel: number analyzed (Participants) | 184
  Fourth Line: Docetaxel | 5
  Fourth Line: Enzalutamide: number analyzed (Participants) | 184
  Fourth Line: Enzalutamide | 11
  Fourth Line: Radium-223: number analyzed (Participants) | 184
  Fourth Line: Radium-223 | 5
  Fourth Line: Other: number analyzed (Participants) | 184
  Fourth Line: Other | 5
  Fourth Line: EOF: number analyzed (Participants) | 184
  Fourth Line: EOF | 14
  Fourth Line: Death: number analyzed (Participants) | 184
  Fourth Line: Death | 71
  Fifth Line: Palliative care: number analyzed (Participants) | 99
  Fifth Line: Palliative care | 27
  Fifth Line: Cabazitaxel: number analyzed (Participants) | 99
  Fifth Line: Cabazitaxel | 6
  Fifth Line: Other: number analyzed (Participants) | 99
  Fifth Line: Other | 12
  Fifth Line: EOF: number analyzed (Participants) | 99
  Fifth Line: EOF | 9
  Fifth Line: Death: number analyzed (Participants) | 99
  Fifth Line: Death | 45

22. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from index until death (event) or end of study identification 31-Dec-2022 (censoring event). Kaplan-Meier method was used for analysis. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: as for outcome 4
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Number of Participants Analyzed' signifies participants evaluable at specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 795 | 558
Months
  Treated Participants: number analyzed (Participants) | 668 | 536
  Treated Participants | 52.6 [47.1 to 63.7] | 27.6 [24.1 to 30.7]
  Untreated Participants: number analyzed (Participants) | 127 | 22
  Untreated Participants | 12.2 [6.5 to 20.0] | 4.2 [1.2 to 9.3]

23. Primary Outcome: Time to Next Treatment (TTNT)
Description: TTNT was defined as time from initiation of the current treatment line until the initiation of the next treatment line (event), death (event), or end of study identification 31-Dec-2022 (censoring event). Data for first, second, third, fourth and fifth line treatment line was provided in this outcome measure. Kaplan-Meier method was used for analysis.
Time Frame: From initiation of current treatment line until initiation of next treatment line, death censoring event, whichever occurred first, maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 644 | 536
Months
  First Line | 9.9 [8.2 to 13.2] | 10.3 [8.4 to 12.1]
  Second Line: number analyzed (Participants) | 285 | 337
  Second Line | 33.1 [18.9 to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with events. | 6.6 [5.5 to 7.7]
  Third Line: number analyzed (Participants) | 58 | 184
  Third Line | NA [NA to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with events. | 4.0 [3.4 to 5.1]
  Fourth Line: number analyzed (Participants) | 58 | 99
  Fourth Line | NA [NA to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with events. | 4.1 [3.1 to 5.3]
  Fifth Line: number analyzed (Participants) | 0 | 45
  Fifth Line |  | NA [NA to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with events.

24. Primary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as time from mCSPC index until mCRPC index (event), death (competing event) or end of study identification period (31-December-2022; censoring event). Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: From mCSPC index until mCRPC index, death or censoring event, whichever occurred first, maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Analysis excluded participants with missing data. Only reporting arm "Participants Diagnosed With mCSPC" is reported as this outcome measure was to be analyzed for participants who had mCSPC and they progressed to mCRPC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Diagnosed With mCSPC
Number analyzed (Participants) | 270
Months | 19.4 [17.3 to 22.0]

25. Primary Outcome: Number of Participants Per Factors Associated With Disease Progression to Castration Resistant
Description: Factors associated with disease progression to castration resistant included age, CCI, De nova mPC and Gleason score. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: From mCSPC index until mCRPC index, death or censoring event, whichever occurred first, maximum up to 24 months; retrospective available data evaluated in this study for approximately 14 months
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With mCSPC
Number analyzed (Participants) | 257
Participants
  Age: 70 to 80 | 101
  Age: >80 | 45
  Age: <70 | 111
  CCI: 0 | 186
  CCI: 1 | 42
  CCI: 2+ | 29
  De novo mPC: No | 77
  De novo mPC: Yes | 180
  Gleason score: 3 to 6 | 7
  Gleason score: 7 | 27
  Gleason score: 8 | 35
  Gleason score: 9 to 10 | 188

26. Primary Outcome: Annual Incidence of mPC, mCSPC and mCRPC
Description: Incidence was calculated by dividing the number of incident participants each year (2014-2022) by the yearly size of background population in PHD. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC). In this outcome measure for arms mCSPC and mCRPC only those participants are reported who were classified or recorded as mCSPC and mCRPC in specified year. All participants reported under Overall Cohort mPC might not have been recognized/classified/recorded as mCSPC and mCRPC for the specified year, hence sum of participants reported against mCSPC and mCRPC might be less than the participants reported for mPC for that specified year.
Time Frame: as for outcome 4
Population: Analysis population: eligible participants whose data were included, observed for evaluation. Here,'Number Analyzed'=participants evaluable for specified rows,for 'Participants Diagnosed with mCRPC' arm for 'untreated' categories for each year = '0' as number of untreated participants were less, when distributed across specified years = <5. According to Findata guidelines, results having <5 participants with events cannot be exported from Findata servers due to participant privacy restrictions.
Measure: Number; unit: Number of new cases per 1000 person year
Groups:
- Participants With mPC: Eligible participants with mPC and whose data were evaluated retrospectively.
Arm/Group | Participants With mPC | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 1083 | 795 | 558
Number of new cases per 1000 person year
  2014: Treated: number analyzed (Participants) | 85 | 53 | 29
  2014: Treated | 16.81 | 10.48 | 5.73
  2014: Untreated: number analyzed (Participants) | 13 | 15 | 0
  2014: Untreated | 2.57 | 2.97 |
  2015: Treated: number analyzed (Participants) | 92 | 64 | 41
  2015: Treated | 18.09 | 12.59 | 8.06
  2015: Untreated: number analyzed (Participants) | 13 | 12 | 0
  2015: Untreated | 2.56 | 2.36 |
  2016: Treated: number analyzed (Participants) | 105 | 61 | 53
  2016: Treated | 20.52 | 11.92 | 10.36
  2016: Untreated: number analyzed (Participants) | 16 | 18 | 0
  2016: Untreated | 3.13 | 3.52 |
  2017: Treated: number analyzed (Participants) | 97 | 64 | 65
  2017: Treated | 18.86 | 12.44 | 12.64
  2017: Untreated: number analyzed (Participants) | 9 | 11 | 0
  2017: Untreated | 1.75 | 2.14 |
  2018: Treated: number analyzed (Participants) | 98 | 60 | 59
  2018: Treated | 18.94 | 11.6 | 11.4
  2018: Untreated: number analyzed (Participants) | 16 | 18 | 0
  2018: Untreated | 3.09 | 3.48 |
  2019: Treated: number analyzed (Participants) | 114 | 84 | 69
  2019: Treated | 21.93 | 16.16 | 13.27
  2019: Untreated: number analyzed (Participants) | 17 | 14 | 0
  2019: Untreated | 3.27 | 2.69 |
  2020: Treated: number analyzed (Participants) | 147 | 106 | 81
  2020: Treated | 28.12 | 20.27 | 15.49
  2020: Untreated: number analyzed (Participants) | 10 | 8 | 0
  2020: Untreated | 1.91 | 1.53 |
  2021: Treated: number analyzed (Participants) | 110 | 85 | 76
  2021: Treated | 20.85 | 16.11 | 14.41
  2021: Untreated: number analyzed (Participants) | 14 | 12 | 0
  2021: Untreated | 2.65 | 2.27 |
  2022: Treated: number analyzed (Participants) | 106 | 91 | 59
  2022: Treated | 19.9 | 17.08 | 11.08
  2022: Untreated: number analyzed (Participants) | 21 | 19 | 0
  2022: Untreated | 3.94 | 3.57 |

27. Primary Outcome: Number of Events Per Participant Year for Outpatient Clinic Contacts, Hospitalization Contacts
Description: Number of events per participant year for outpatient clinic contacts, hospitalization contacts were reported in this outcome measure. Index date for (i) mCSPC participants were defined as date for the first record of mPC (ii) mCRPC participants were defined as date for progression to castration resistant (if =3 months from castration-sensitive treatment initiation [1st control usually at 3 months], considered de novo CRPC).
Time Frame: From index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx. 9 years; retrospective available data evaluated in this study for approximately 14 months
Population: Analysis population included all eligible participants whose data were included and observed for evaluation in the study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Events per participant per year
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 668 | 532
Events per participant per year
  Outpatient Clinic Contacts | 14.2 [13.2 to 15.4] | 18.6 [17.3 to 20.1]
  Hospitalization Contacts | 0.7 [0.6 to 0.7] | 1.2 [1.0 to 1.3]

28. Primary Outcome: Number of Days Per Participant Year for Hospital Inpatient Days
Description: Number of days per participant year for hospital inpatient days were reported in this outcome measure.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Mean (95% Confidence Interval); unit: Days per participant year
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
Number analyzed (Participants) | 668 | 532
Days per participant year | 3.1 [2.6 to 3.6] | 6.5 [5.7 to 7.4]

ADVERSE EVENTS:
Time Frame: All-cause mortality: from index date to end of follow-up date [death or end of identification 31-Dec-2022, whichever occurred first], maximum up to approx.9 years; retrospective available data evaluated in this study for approximately 14 months; for adverse events time frame was not applicable as they were not assessed in this study
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (that is, identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events (serious and other) were not planned to be evaluated and at risk is "0".
Arm/Group | Participants Diagnosed With mCSPC | Participants Diagnosed With mCRPC
All-Cause Mortality (participants affected / at risk) | 343/795 | 218/558
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT05701007/Prot_SAP_000.pdf